CLINICAL TRIAL: NCT02939079
Title: Evaluating the Effect of Fingolimod With Fish Oil Compared to Fingolimod With Placebo on Tumor Necrosis Factor-α , Interleukin1b , Interleukin6, and Interferon-gamma in Patients With Relapsing-Remitting Multiple Sclerosis
Brief Title: Evaluating of the Effect of Fingolimod With Fish Oil on Relapsing-Remitting Multiple Sclerosis Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Vahid Shaygannejad, Associate Professor of Neurology, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 293396
Record Dates: First submitted 2016-10-14; First posted 2016-10-19 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Fingolimod; Fish Oil
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fingolimod and Fish Oil (Experimental): Fingolimod 0.5 mg capsule daily by mouth and Fish Oil 1 g capsule daily by mouth for one year.
  Interventions: Drug: Fingolimod; Dietary Supplement: Fish Oil
- Fingolimod and Placebo (Active Comparator): Fingolimod 0.5 mg capsule daily by mouth and Placebo capsule daily by mouth for one year.
  Interventions: Drug: Fingolimod; Drug: Placebo (for Fish Oil)

INTERVENTIONS:
Drug: Fingolimod — Produced by Osveh ® Pharm Company in Iran
  Other Names: Fingolid ®
Dietary Supplement: Fish Oil — produced by Zahravi ® Pharm Company in Iran
  Other Names: CODLIVE ®; OMEGAMAX ®
  Arms: Fingolimod and Fish Oil
Drug: Placebo (for Fish Oil) — placebo capsules to mimic Fish Oil 1 g capsules
  Arms: Fingolimod and Placebo

SUMMARY:
This study evaluates the effect of adding fish oil to Fingolimod on some serum cytokines in patients with Relapsing-Remitting Multiple Sclerosis.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic autoimmune disease characterized by inflammatory demyelinative lesions in central nervous system. Relapsing-Remitting MS is the most common form of the disease observed in 85% of patients. This form presents with acute or sub-acute onset of neurological symptoms and patients may fully or partially recover and relapses may occur from time to time.

Regarding MS pathogenesis, the findings suggest the role of environmental factors in triggering the innate immune system and activating T cells and the onset of a chronic inflammatory response against myelin antigens in the central nervous system in people who are genetically prone to the disease. Among immune cells, T helper 17 (Th17) plays an important role in autoimmune response and are shown to be involved in clinical course of Relapsing-Remitting MS. Th17 cell differentiation is controlled by several cytokines, including interleukin-6 (IL-6), interleukin-1b (IL-1b) and interleukin-10 (IL-10). Also, IL 6 have an inhibitory effect on Th17 cell differentiation through increased production of interferon-gamma (IFN-gamma) and IL 10.

Currently, immunomodulatory drugs are considered as the first line treatment in MS. Fingolimod is the first oral immunomodulatory medication used for Relapsing-Remitting MS. It is phosphorylated by crossing the blood-brain barrier and is converted to its active metabolite, Fingolimod-P. This metabolite acts as a Sphingosine-1-phosphate receptor (S1PR1) on oligodendrocytes, microglias, astrocytes, and neurons and inhibits the entry of lymphocytes into the central nervous system. Therefore, it reduces demyelination and may also lead to remyelination.

Nutrition is known as a possible environmental factor in pathogenesis of MS. Positive clinical and biological effects of dietary supplements containing polyunsaturated fatty acids omega -3 (PUFA) in the course of autoimmune diseases such as MS have been studied. High levels of PUFA is found in fish oil which is also known as an antioxidant, anti-inflammatory and immunomodulatory agent. Several studies have evaluated the effect of fish oil as a dietary supplement in the treatment of MS however, conflicting findings are reported.

In this study, the investigators aim to evaluate the effect of Fingolimod with Fish oil compared to Fingolimod with placebo on TNF-α, IL1b, IL6, and IFN-gamma in patients with Relapsing-Remitting Multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing-remitting multiple sclerosis according to McDonald's criteria (2010)
* Age between 18 and 45 years
* Expanded Disability Status Scale (EDSS) between 0-5
* History of at least one relapse during the last year
* Intolerance or serious complications when receiving interferons
* Not receiving interferons in the last two months
* Not having relapse in the last 30 days
* Negative pregnancy test
* History of varicella or varicella vaccination, or positive test for anti-varicella antibodies
* Not to take any medication or dietary complement without permission of the physician
* Filling informed consent

Exclusion Criteria:

* Having chronic and infectious diseases
* History of cardiovascular diseases
* Taking corticosteroids in the last 30 days
* Taking chemotherapy agents such as Cyclophosphamide
* Patients who have taken fingolimod before
* Patients who experience relapse during the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaygannejad Shaygannejad, M.D., Study Chair — Isfahan University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided
The investigators may make individual participant data available regarding drug side effects or other factors that need to be described individually however the primary outcome will be published as group result and not individual results.

REFERENCES:
- [Background] Aktas O, Kury P, Kieseier B, Hartung HP. Fingolimod is a potential novel therapy for multiple sclerosis. Nat Rev Neurol. 2010 Jul;6(7):373-82. doi: 10.1038/nrneurol.2010.76. Epub 2010 Jun 15. PMID 20551946
- [Background] Brinkmann V, Billich A, Baumruker T, Heining P, Schmouder R, Francis G, Aradhye S, Burtin P. Fingolimod (FTY720): discovery and development of an oral drug to treat multiple sclerosis. Nat Rev Drug Discov. 2010 Nov;9(11):883-97. doi: 10.1038/nrd3248. Epub 2010 Oct 29. PMID 21031003
- [Background] Gallai V, Sarchielli P, Trequattrini A, Franceschini M, Floridi A, Firenze C, Alberti A, Di Benedetto D, Stragliotto E. Cytokine secretion and eicosanoid production in the peripheral blood mononuclear cells of MS patients undergoing dietary supplementation with n-3 polyunsaturated fatty acids. J Neuroimmunol. 1995 Feb;56(2):143-53. doi: 10.1016/0165-5728(94)00140-j. PMID 7860710
- [Background] Kappos L, Radue EW, O'Connor P, Polman C, Hohlfeld R, Calabresi P, Selmaj K, Agoropoulou C, Leyk M, Zhang-Auberson L, Burtin P; FREEDOMS Study Group. A placebo-controlled trial of oral fingolimod in relapsing multiple sclerosis. N Engl J Med. 2010 Feb 4;362(5):387-401. doi: 10.1056/NEJMoa0909494. Epub 2010 Jan 20. PMID 20089952
- [Background] Nordvik I, Myhr KM, Nyland H, Bjerve KS. Effect of dietary advice and n-3 supplementation in newly diagnosed MS patients. Acta Neurol Scand. 2000 Sep;102(3):143-9. doi: 10.1034/j.1600-0404.2000.102003143.x. PMID 10987373
- [Background] Ramirez-Ramirez V, Macias-Islas MA, Ortiz GG, Pacheco-Moises F, Torres-Sanchez ED, Sorto-Gomez TE, Cruz-Ramos JA, Orozco-Avina G, Celis de la Rosa AJ. Efficacy of fish oil on serum of TNF alpha , IL-1 beta , and IL-6 oxidative stress markers in multiple sclerosis treated with interferon beta-1b. Oxid Med Cell Longev. 2013;2013:709493. doi: 10.1155/2013/709493. Epub 2013 Jun 18. PMID 23861993
- [Background] Torkildsen O, Wergeland S, Bakke S, Beiske AG, Bjerve KS, Hovdal H, Midgard R, Lilleas F, Pedersen T, Bjornara B, Dalene F, Kleveland G, Schepel J, Olsen IC, Myhr KM. omega-3 fatty acid treatment in multiple sclerosis (OFAMS Study): a randomized, double-blind, placebo-controlled trial. Arch Neurol. 2012 Aug;69(8):1044-51. doi: 10.1001/archneurol.2012.283. PMID 22507886

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period started on April 2015. 74 patients were screened initially and 50 of them were recruited. All the patients were recruited from the neurology department of Kashani hospital, Isfahan, iran. They were patients referred to the neurology department (multiple sclerosis clinic) for evaluation and treatment.
Pre-assignment Details: After recruitment, no medication was prescribed for the patients for two months as the wash-out period. Then patients were assigned to study groups.
Period: Overall Study
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Started | 25 | 25
Completed | 21 | 20
Not Completed | 4 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — relapse during the study | 1 | 1

BASELINE CHARACTERISTICS:
Population: We used a per-protocol analysis approach.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.19 (9.97) | 31.40 (8.41) | 33.34 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 8 | 4 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Iran | 21 | 20 | 41
Dietary habits, Categorical (seafood meals per month) [Count of Participants; unit: Participants]
  0-1 meals per month | 19 | 18 | 37
  2-4 meals per month | 2 | 2 | 4
  >4 meals per month | 0 | 0 | 0
EDSS [Mean (Standard Deviation); unit: units on a scale] — Expanded disability status scale (EDSS) is a measure of disability for patients. The score ranges from 0-10, with 0 showing normal neurological exam and 10 showing death due to the disabling disease. Thus, higher scores represent more profound levels of disability.
  units on a scale | 3.10 (1.28) | 2.55 (1.38) | 2.83 (1.33)

OUTCOME MEASURES:

1. Primary Outcome: Serum Level of TNF-α
Description: 5 cc of venous blood is taken from patients and are kept in test tubes without ethylenediaminetetraacetic acid (EDTA). Test tubes are kept one hour immobilized so that clotted blood and serum are separated. Then, the serum is divided into four samples of 0.5 cc for immunologic testing of all primary outcomes. Immunologic testing is performed by sandwich ELISA method using Diaclone ® kits (made in France) and according to manufacturer's instructions.
Time Frame: Baseline
Population: Per-protocol analysis
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 37.16 (92.74) | 28.79 (47.46)

2. Primary Outcome: Serum Level of IL1b
Description: 5 cc of venous blood is taken from patients and are kept in test tubes without EDTA. Test tubes are kept one hour immobilized so that clotted blood and serum are separated. Then, the serum is divided into four samples of 0.5 cc for immunologic testing of all primary outcomes. Immunologic testing is performed by sandwich ELISA method using Diaclone ® kits (made in France) and according to manufacturer's instructions.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 13.76 (0.74) | 14 (1.03)

3. Primary Outcome: Serum Level of IL6
Description: as for outcome 2
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 6.19 (0.35) | 6.33 (0.58)

4. Primary Outcome: Serum Level of IFN-gamma
Description: as for outcome 2
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 6.38 (1.51) | 6.98 (3.87)

5. Primary Outcome: Serum Level of TNF-α
Description: as for outcome 2
Time Frame: 6 months after intervention
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 28.03 (60.36) | 17.18 (18.88)

6. Primary Outcome: Serum Level of TNF-α
Description: as for outcome 2
Time Frame: 1 year after intervention
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 21.20 (36.45) | 16.47 (16.64)

7. Primary Outcome: Serum Level of IL1b
Description: as for outcome 2
Time Frame: 6 months after intervention
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 13.61 (0.58) | 13.47 (0.74)

8. Primary Outcome: Serum Level of IL1b
Description: as for outcome 2
Time Frame: 1 year after intervention
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 13.17 (0.52) | 13.15 (0.61)

9. Primary Outcome: Serum Level of IL6
Description: as for outcome 2
Time Frame: 6 months after intervention
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 6.65 (2.11) | 6.17 (0.71)

10. Primary Outcome: Serum Level of IL6
Description: as for outcome 2
Time Frame: 1 year after intervention
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 6.17 (0.76) | 6.05 (0.47)

11. Primary Outcome: Serum Level of IFN-gamma
Description: as for outcome 2
Time Frame: 6 months after intervention
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 5.71 (0.57) | 6.37 (1.77)

12. Primary Outcome: Serum Level of IFN-gamma
Description: as for outcome 2
Time Frame: 1 year after intervention
Measure: Mean (Standard Deviation); unit: Pg/ml
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
Number analyzed (Participants) | 21 | 20
Pg/ml | 5.92 (1.31) | 5.99 (0.84)

ADVERSE EVENTS:
Time Frame: Patients were evaluated in the study for one year and were observed for adverse events during this period.
Description: Adverse events were collected through follow up phone calls and visits.
Arm/Group | Fingolimod and Fish Oil | Fingolimod and Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25 | 2/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fingolimod and Fish Oil (N=25) | Fingolimod and Placebo (N=25)
Hypotension and bradycardia (Cardiac disorders) | 2 (2) | 2 (2) — Adverse effects stopped after medication discontinuation in all cases.

LIMITATIONS AND CAVEATS:
Small sample size and trial duration; Not giving patients specific nutritional diets; Receiving tocopherol in the placebo capsules which may confound our findings considering the antioxidant nature of tocopherol; Lower doses of fish oil prescribed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes